CLINICAL TRIAL: NCT02895191
Title: A Randomized, Blind, Placebo-controlled, Parallel Group, Multi-center Study to Evaluate the Safety and Dose Response Relationship of Ulinastatin for Acute Respiratory Distress Syndrome(ARDS)
Brief Title: The Safety and Dose Response Relationship of Ulinastatin for Acute Respiratory Distress Syndrome(ARDS)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Techpool Bio-Pharma Co., Ltd. (Industry)
Collaborators: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UTI-2001
Record Dates: First submitted 2016-07-21; First posted 2016-09-09 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — urinastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 (Experimental): Cohort 1- Ulinastatin 4.8 million units per day
  Interventions: Drug: ulinastatin
- Cohort 2 (Experimental): Cohort 2- Ulinastatin 2.4 million units per day
  Interventions: Drug: ulinastatin
- Cohort 3 (Experimental): Cohort 3- Ulinastatin 1.2 million units per day
  Interventions: Drug: ulinastatin
- control group (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ulinastatin — Patients will receive the study drugs for 7 to 14 days
  Other Names: UTI; urinary trypsin inhibitor; bikunin
  Arms: Cohort 1; Cohort 2; Cohort 3
Drug: placebo — Patients will receive the placebo for 7 to 14 days
  Arms: control group

SUMMARY:
Compared with placebo, evaluate the effects and safety of Ulinastatin(UTI) added to conventional treatment for ARDS; Evaluate the dose response relationship of Ulinastatin for ARDS.

DETAILED DESCRIPTION:
After signed off the informed consent form by patient or surrogate, and after completing the screening phase, the patients who fulfill the inclusion and exclusion criteria will be randomized 1:1:1:1 to the 4 study arms. All the Patients will receive the study treatment drugs for 7 to 14 days. Use Day 28 of last patient as a cut-off day, Collect the follow up visit data on both Day 28 and Day 90 of other patients．

ELIGIBILITY:
Inclusion Criteria:

1. Have provided signed written informed consent form (ICF) from the patient or the patient's legal representative;
2. Male or Female patients ≥18 years of age;
3. ARDS defined with using 2012 Berlin Criteria;
4. ARDS diagnosed ≤7 days, and patients should be mechanically ventilated(invasive and or noninvasive mechanical ventilation); 5)100mmhg < PaO2/FiO2 < 250mmhg with CPAP/PEEP≥5 cmH2O;

Exclusion Criteria:

1. Patient with known hypersensitivity to Ulinastatin/adjuvant or patient with allergic constitution;
2. Patients with artificial organs replacement therapy for liver or kidney；
3. Glasgow Coma Scale (GCS)≤8；
4. Cardiogenic pulmonary edema , and the cardiogenic pulmonary edema is as the only or primary reason for respiratory failure;
5. ARDS caused by burning, drowning, poisoning;
6. Presence of severe chronic liver diseases (Child-Pugh score 12-15)，or severe chronic respiratory disease with a PaCO2 > 50 mmHg or the use of home oxygen;
7. Neutrophils<1.5×10^9/L
8. Moribund patients (i.e.,expected to live no longer than 24 hours) or with recent (within 7days or anytime during present hospitalization) cardiopulmonary arrest;
9. Patients need long-term glucocorticoid treatment or need to be treated with immunosuppressive drugs;
10. No intent/unwillingness to follow lung protective ventilation strategy or fluid management protocol;
11. Lung transplant patients;
12. Patients with malignancy, expected to live no longer than 6 months;
13. Pregnant or breast-feeding;
14. Patients who have participated in any clinical study within 3 months prior to the screening;
15. Any condition that in the opinion of the investigator would add the patient's risk or jeopardize the operation of the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse events(AEs) which can not excluded relatedness with study Product | Day 1 to Day 90

SECONDARY OUTCOMES:
Changes of PaO2/FiO2 ratio | Day 0 and Day 1 to within 24h after the last treatment
Days alive and off ventilator | Day 1 to Day 28
Days in the ICU | Day 1 to Day 14
Changes of pulmonary compliance | Day 1 , Day 3 ,Day7 and within 24h after the last treatment
Rate of new organ failure | Day 1 to Day 90
Changes of APACHEⅡ Score from baseline | Day 3 ,Day7 and within 24h after the last treatment
Changes of Murray Lung Injury Score from baseline | Day 3 ,Day7 and within 24h after the last treatment
Changes of Sequential Organ Failure Assessment (SOFA) score from baseline | Day 3 ,Day7 and within 24h after the last treatment
All-cause mortality | Day 28 , Day 90 and Day 1 to Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Yimin Li, Doctor, Principal Investigator — First Affiliated Hospital of Guangzhou Medical University
Locations (11):
- China (11):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Hainan General Hospital, Haikou, Hainan
  - Huadong Hospital,Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital, Shanghai, Shanghia
  - West China Hospital,Sichuan Unversity, Chengdu, Sichuan
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Zhejiang Hospital, Hangzhou, Zhejiang
  - Lishui City People's Hospital, Lishui, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided